CLINICAL TRIAL: NCT02234206
Title: Safety and Efficacy of Chandrakanthi Choornam in Oligospermia - A Preclinical and Clinical Study
Brief Title: A Clinical Trial to Study the Safety and Efficacy of Chandrakanthi Choornam in Patients With Low Sperm Count
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Responsible Party: Principal Investigator, Dr.B.Akila., M.D (s), Safety and Efficacy of Chandrakanthi Choornam in Oligospermia - A Preclinical and Clinical Study, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ref.No. ExII(1)/29096/2011; CTRI/2014/01/004281 (Registry Identifier: CLINICAL TRIALS REGISTRY- INDIA)
Record Dates: First submitted 2014-08-27; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Oligospermia
Keywords: Hypospermatogenesis, Low Sperm Count, Oligozoospermia
MeSH Terms: conditions — Oligospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chandrakanthi choornam (Experimental): Chandrakanthi Choornam (CKC) - 12gm in milk
  OD dose; Oral route
  3 Months - duration
  Intervention Drug: Chandrakanthi Choornam (CKC)
  Interventions: Drug: Chandrakanthi Choornam (CKC)

INTERVENTIONS:
Drug: Chandrakanthi Choornam (CKC) — 12gm in milk - OD dose; Oral route; 3 Months ( 90days) - duration
  Preparation from approved sastric book as per drugs & cosmetic act 1940
  Other Names: Nerunjil choornam

SUMMARY:
This is an Open clinical trial to study the safety and efficacy of Chandrakanthi Choornam in 40 patients with Oligospermia. Chandrakanthi choornam is a formulation consisting of 25 ingredients. They are Curculigo orchioides -rhizome, Madhuca longifolia - flower, Cinnamomum verum -bark,Cinnamomum tamala-Leaf, Syzygium aromaticum - flower bud,Coscinium fenestratum-stem bark,Mesua ferrea-flower, Maerua arenaria-tuber, Adhatoda vasica- seed, Moringa oleifera-seed, Lawsonia inermis-seed, Vitis vinifera- fruit, Bombax ceiba- gum, Bambusa aurundinaceae-salt,Phoenix dactilifera- fruit,Ilicium verum- flower, Mucuna prurita-seed, Cyperus rotundus- rhizome, Glycyrrhiza glabra-root, Tribulus terrestris-fruit, Cuminum cyminum-seed,Costus speciosus-root,Myrsitica fragrans-seed, Alternanthera sessilis-seed and asphaltum-mineral. Treatment duration is three months.Study is conducted in India (Chennai). Primary outcome measure is to see the changes in sperm count, motility and morphology. Secondary Outcome measure is to see the impact on the harmone level.

DETAILED DESCRIPTION:
METHODOLOGY OF PROPOSED RESEARCH:

I. Preclinical study II. Clinical study

I. PRECLINICAL STUDY:

Standardization Of The Study Drug

1. Botanical Identification
2. Chemical Identification
3. Preparation of the study drugs:

   Formulation: Chandrakanthi choornam Source : Chikicharathna deepam Part II. Pg-168 (Approved sastric book as per drugs & cosmetic act 1940.
4. Chemical methods of testing
5. Pharmacological study : A. Spermotogenic Activity
6. Toxicological study : A. Acute Toxicity B. Long term Toxicity

II. CLINICAL STUDY

Conducted as per the guidelines of GCP accepted by Ayush adapted from the ICH.

A. Pilot study B. Main study

ELIGIBILITY:
Inclusion criteria:

* Male infertile Patients with age between 21-45 yrs
* Marriage history for >1 year
* Abnormal Sperm count 1-15 million/ml
* Patients with normal Liver & Renal function test
* Willing to give specimen of semen before & at the end of the clinical trial
* Informed patients giving written consent

Exclusion criteria:

* Azoospermia - complete absence of sperm cells in the ejaculate
* Aspermia - complete lack of semen
* Necrospermia- Spermatozoa in semen are either immobile or dead.
* Clinical diagnosis of Varicocele & Hydrocele
* History of Undescended testis
* Inguinal hernia on physical examination
* Male accessory gland infection
* History of DM, Hypertension and Cardiac disease
* Any recent medical or surgical illness
* Underwent treatment for promoting Spermatogenic fertility in last 3 months
* Other Systemic disease requiring specific therapies
* Known Thyroid disease
* Past history of Renal, Hepatic or any other chronic illness in the Patient

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sperm concentration per milliliter of seminal fluid | 90 days
  Changes in the total number of sperm cells per milliliter of seminal fluid were evaluated from baseline to three months
Proportion of Sperm motility | 90 days
  Changes in the percentage of total and progressive motility of sperm were evaluated from baseline to three months
Proportion of Sperm morphology | 90 days
  Changes in the percentage of sperm cells with normal forms were evaluated from baseline to three months

SECONDARY OUTCOMES:
Impact on the hormonal level due to the clinical trial | 90 days
  Changes in serum Testosterone, LH and FSH were estimated from baseline to three months

OTHER OUTCOMES:
Assessment on Safety parameters | 90 days
  Safety parameters: Liver function test ,Renal function test , Lipid profile, Haematological profile , Blood Glucose, Urinary parameters were assessed from baseline to three months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.B. Akila., M.D (s), Principal Investigator — National institute of Siddha
Locations (1):
- National institute of siddha, Chennai, Tamil Nadu, India